CLINICAL TRIAL: NCT04852354
Title: Tissue Collection for Drug Screening and Bioanalysis
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 20-01021289
Record Dates: First submitted 2021-04-10; First posted 2021-04-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Central Nervous System Tumor
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Tumor patients undergoing neurosurgery: Samples of tumor tissue, blood, CSF, saliva, skull, and dura will be taken during neurosurgery from tumor patients meeting the inclusion criteria.
- Parents of tumor patients: Saliva samples will be taken from parents of tumor patients meeting the inclusion criteria.
- Cohort 2: Non-Tumor patients undergoing neurosurgery: Blood and CSF samples will be taken from non-tumor patients meeting the inclusion criteria.
- Cohort 3: Autopsy tumor tissue donation: Post-mortem biospecimens such as whole brain, spinal cord, biofluids (e.g., cerebrospinal fluid and blood) and skin biopsy will be collected through autopsy donation from brain tumor patients meeting the inclusion criteria.

SUMMARY:
The purpose of this study is to improve upon the knowledge currently available about central nervous system (CNS) tumors. We will study the different characteristics of these tumors using tissue samples collected during surgery and post-autopsy. The aim is to create tumor cell lines and models to test how they respond to different drugs. This research will help improve treatment options and identify new targets for therapy.

DETAILED DESCRIPTION:
The goal of this project is to enable the acquisition of tissue available for research with the prospect of enabling the development of new therapeutic avenues for patients diagnosed with cancer in the central nervous system.

During patients' (with a CNS tumor) routine operative procedure, if extra tissue deemed unnecessary for diagnostic or clinical purposes is available, selected samples will undergo DNA and/or RNA extraction and integrity analysis, whole genome and RNA sequencing, DNA and RNA methylome analyses, proteomic analysis, immunoprofiling, and primary culturing of the tumor cells. These cultures may then be used for drug screenings and to create patient-derived xenografts, or for comparisons between tumor and non-tumor patients. Other biological samples may be collected. Tissue collection for drug screening will be extended to post-mortem biospecimens such as whole brain, spinal cord, biofluids (e.g., cerebrospinal fluid and blood) and skin biopsy. These samples will be collected through autopsy donation from pediatric and adult brain tumor patients.

Additionally, saliva samples may be obtained from the parents of pediatric patients with CNS tumors, and biological samples may be collected from pediatric patients without a CNS tumor who are undergoing a neurological procedure. These samples may be used for comparison with samples from patients with CNS tumors.

ELIGIBILITY:
Inclusion Criteria for Tumor patients undergoing neurosurgery (cohort 1)

1. Subject has presented with a suspected/confirmed neoplastic CNS lesion and is undergoing a neurosurgical procedure in which CNS tissue and/or tumors associated with this tissue will be removed.
2. There must be tissue available in excess of that required by neuropathology for diagnostic purposes.
3. Subject of all ages included.
4. Subjects who are pregnant can be included.
5. Subjects who are neonates (0-4 weeks) can be included.

Inclusion Criteria for Non-tumor patients undergoing neurosurgery (cohort 2)

1. Subject is between 4 weeks and 21 years of age and is undergoing a neurosurgical procedure at WCMC.
2. Subject does not have a CNS tumor diagnosis.
3. Subject should not be pregnant at the time of enrollment.

Inclusion Criteria for Autopsy tumor tissue donation (cohort 3)

1. Subject of all ages included
2. Subject has been diagnosed with a neoplastic CNS lesion at the time of passing.
3. Subjects who are pregnant can be included.
4. Subjects who are neonates (0-4 weeks) can be included.

Inclusion Criteria for parent of tumor patients

1. Subject is the biological parent of a patient undergoing/ who underwent a neurosurgical procedure in which CNS tissue and/or tumors associated with this tissue will be/ was removed.
2. Subject is the biological parent of patient enrolled in cohort 1.
3. Subject is not pregnant at the time of enrollment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a central nervous system tumors. Parents of patients with CNS tumors.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2029-07-22 (Estimated); Study Completion 2029-07-22 (Estimated)

PRIMARY OUTCOMES:
Evaluating and characterizing the genetic, immunohistochemical, cellular, and molecular profiles of pediatric neoplastic lesions | Through study completion, average 1-3 years
  To develop patient-derived tissue cell lines and xenografts

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Greenfield, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajappa P, Cobb WS, Vartanian E, Huang Y, Daly L, Hoffman C, Zhang J, Shen B, Yanowitch R, Garg K, Cisse B, Haddock S, Huse J, Pisapia DJ, Chan TA, Lyden DC, Bromberg JF, Greenfield JP. Malignant Astrocytic Tumor Progression Potentiated by JAK-mediated Recruitment of Myeloid Cells. Clin Cancer Res. 2017 Jun 15;23(12):3109-3119. doi: 10.1158/1078-0432.CCR-16-1508. Epub 2016 Dec 30. PMID 28039266